CLINICAL TRIAL: NCT06848647
Title: Treatment of Sleep Apnea to Improve Metabolic Health - a Novel Approach to Unanswered Questions
Brief Title: Treatment of Sleep Apnea to Improve Metabolic Health
Acronym: GLYCOSACT
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01150-01; 2023-05223-02; 20230298 (Other Grant/Funding Number: Swedish Heart Lung Foundation)
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Sleep Apnea, Obstructive; Metabolism; CPAP; Patients Above 18 Years
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Diabetes and prediabetes prevail among obstructive sleep apnea (OSA) patients. OSA and short sleep both detrimentally affect glycemic control regardless of obesity. With 1 in 10 adults having diabetes, 1 in 10 with prediabetes, and an estimated 600,000 affected by OSA in Sweden, attaining glycemic control is crucial. Though continuous positive airway pressure (CPAP) is the most effective treatment for OSA, its application lacks personalization, ignoring factors like comorbidities and sleep duration. Key unanswered questions regarding CPAP's impact on glycemic control include: 1) Does high CPAP adherence optimize glycemic control? 2) Should short sleep be addressed alongside OSA treatment for glycemic control? 3) Does long-term diabetes hinder CPAP's glycemic control efficacy? The purpose of this project is to enable precision health in CPAP treatment and producing a personalized treatment model for achieving glycemic control in patients with OSA, treated with CPAP. Taking advantage of a large unique patient cohort (600 patients followed over 18 months) with extensive and objective measures on CPAP adherence, OSA reduction, sleep duration, as well as information on comorbidities, anthropometric, lifestyle data, and a wide range of biomarkers related to glycemic control. This comprehensive approach and in-depth analysis will address these questions and generate a personalized treatment strategy for glycemic control in CPAP-treated OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with obstructive sleep apnea
* Planned for CPAP treatment
* 18 years and above

Exclusion Criteria:

* Patient not wanting to participate in study
* Non-Swedish speaking
* Judged by physician as non-fit for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive sleep apnea referred to the Sleep Apnea Unit at Uppsala University Hospital for CPAP treatment
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Homeostatic model assessment for insulin resistance (HOMA-IR) | From enrollment to the end of treatment at 12 months
  Clinical marker: HOMA-IR calculated from blood glucose and serum insuling
Glycated hemoglobin (HbA1c) | From enrollment to the end of treatment at 12 months
  Clinical maker: glycated hemoglobin (HbA1c) in % and mmol/mol
Blood glucose | From enrollment to the end of treatment at 12 months
  Clinical marker: blood glucose in mmol/L
Serum insulin | From enrollment to the end of treatment at 12 months
  Clinical marker: serum insulin in mU/L
Plasma triglycerides | From enrollment to the end of treatment at 12 months
  Clinical marker: Triglycerides in mg/dL
Plasma cholesterol | From enrollment to the end of treatment at 12 months
  Clinical marker: plasma cholesterol in mg/dL
HDL-cholesterol | From enrollment to the end of treatment at 12 months
  Clinial marker: high-density lipoprotein (HDL) cholesterol in mg/dL
LDL-cholesterol | From enrollment to the end of treatment at 12 months
  Clinical marker: low-density lipoprotein (LDL) cholesterol in mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No